CLINICAL TRIAL: NCT02357043
Title: User Performance Evaluation for DARIO™ Blood Glucose Monitoring System (BGMS)
Brief Title: User Performance Evaluation for DARIO™ BGMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LabStyle Innovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP-0002
Record Dates: First submitted 2015-01-21; First posted 2015-02-06 (Estimated); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2016-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dario Blood Glucose Monitoring System (Experimental): Subject will be requested to follow the device instructions and perform his/her own finger-stick test using the Dario Glucose Monitoring System (BGMS).
  Interventions: Device: Dario Blood Glucose Monitoring System; Device: YSI

INTERVENTIONS:
Device: Dario Blood Glucose Monitoring System — Finger-stick obtained with BGMS
Device: YSI — Finger-stick sample obtained by nurse/technician to be tested with YSI

SUMMARY:
The study aims to evaluate the accuracy of the blood glucose level results obtained from fingertip using the Dario Blood Glucose Monitoring System (BGMS) compared to Yellow Springs Instrument (YSI) as well as to evaluate the usability of the Dario Blood Glucose Monitoring System (BGMS) by laypersons using only device labeling.

DETAILED DESCRIPTION:
Each subject enrolled in the study will be requested to follow the device instructions and perform his/her own finger-stick test using the Dario Blood Glucose Monitoring System (BGMS). Immediately after the subject tested him/herself a trained nurse/technician will collect another blood sample from the subject for testing by the Yellow Springs Instrument (YSI). The subject will complete a usability questionnaire on his/her experience using the Dario Blood Glucose Monitoring System (BGMS) and the nurse/technician will complete a questionnaire assessing the subject's performance. A venous blood sample for Complete Blood Count (CBC) will be taken by the nurse/technician and sent for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has Type I or Type II diabetes
2. Subject speaks and reads English proficiently
3. Subjects owns and uses Android and iOS based smart mobile device for at least 1 year
4. Subject is able and agrees to sign the informed consent form (minor subjects must be accompanied by a parent or legal guardian to provide consent for their participation in the study).

Exclusion Criteria:

1. Subject has medical training or works in the field of Blood Glucose Monitoring System (BGMS)
2. Subject is critically ill
3. Subject has an impairment that prevents him/her to follow the study procedures
4. Subject has any condition that the Principal Investigator believes may interfere in the subject's participation in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Remington-Davis, Inc., Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dario Blood Glucose Monitoring System
Started | 368
Completed | 368
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dario Blood Glucose Monitoring System
Number analyzed (Participants) | 368
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 300
  >=65 years | 65
Age, Continuous [Mean (Full Range); unit: years] | 52.4 [13 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 199
Race/Ethnicity, Customized [Number; unit: participants]
  Americam Indian or Alaska Natice | 3
  Asian | 7
  Black or African America | 81
  Hispanic or Latino | 1
  Native Hawaiian or other Pacific Ilander | 1
  White | 267
  Other | 8
Region of Enrollment [Number; unit: participants]
  United States | 368

OUTCOME MEASURES:

1. Primary Outcome: Accuracy - Blood Glucose Level Obtained by Layperson With the Dario Meter Compared to Blood Glucose Level on Yellow Springs Instrument Obtained by Nurse/Technician
Description: Blood Glucose Level obtained by layperson on Dario meter versus Blood Glucose Level by Yellow Springs Instrument (obtained by nurse/technician)
Time Frame: 5 minutes
Measure: Number; unit: Participants
Arm/Group | Dario Blood Glucose Monitoring System
Number analyzed (Participants) | 368
Participants
  < 75 mg/dl Within ±5mg/dL | 12
  < 75 mg/dl Within ±10mg/dL | 22
  < 75 mg/dl Within ±15mg/dL | 24
  >=75 mg/dl Within ±5% | 134
  >=75 mg/dl Within ±10% | 257
  >=75 mg/dl Within ±15% | 328
  >=75 mg/dl Within ±20% | 339
  < 100 mg/dl Within ±5mg/dL | 42
  < 100 mg/dl Within ±10mg/dL | 73
  < 100 mg/dl Within ±15mg/dL | 91
  >= 100 mg/dl Within ±5% | 111
  >= 100 mg/dl Within ±10% | 211
  >= 100 mg/dl Within ±15% | 265

ADVERSE EVENTS:
Arm/Group | Dario Blood Glucose Monitoring System
Serious Adverse Events (participants affected / at risk) | 0/368
Other Adverse Events (participants affected / at risk) | 0/368

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days